CLINICAL TRIAL: NCT06723964
Title: A Phase 1 Dose-Escalation Study to Evaluate the Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of AP505 Injection, an Anti-PD-L1 and Anti-VEGF Bispecific Antibody, in Patients With Advanced Solid Tumors
Brief Title: A Study of AP505 Injection in Patients With Advanced Malignant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AP Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP505-101
Record Dates: First submitted 2024-11-22; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- AP505 0.035 mg/kg (Experimental): AP505 0.035 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 0.12 mg/kg (Experimental): AP505 0.12 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 0.4 mg/kg (Experimental): AP505 0.4 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 1.2 mg/kg (Experimental): AP505 1.2 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 4.0 mg/kg (Experimental): AP505 4.0 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 8.0 mg/kg (Experimental): AP505 8.0 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 11.0 mg/kg (Experimental): AP505 11.0 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 15.0 mg/kg (Experimental): AP505 15.0 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 20.0 mg/kg (Experimental): AP505 20.0 mg/kg Open Label
  Interventions: Drug: AP505
- AP505 25.0 mg/kg (Experimental): AP505 25.0 mg/kg Open Label
  Interventions: Drug: AP505

INTERVENTIONS:
Drug: AP505 — AP505 is a Anti-PD-L1 and Anti-VEGF Antibody Fusion Protein.

SUMMARY:
This is a multi-center, open-label study to investigate the safety, tolerability, pharmacokinetics (PK), immunogenicity, and preliminary anti-tumor activity of AP505 injection in patients with advanced solid tumors. The study will determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) for AP505.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet ALL of the inclusion criteria described.

1. Voluntarily participate in this study and provide a signed and dated informed consent form (ICF).
2. Male or female aged ≥ 18 years old (inclusive) at the time of signing the ICF.
3. Patients with histologically and/or cytologically confirmed advanced solid tumor, who have failed established standard medical anti-cancer therapies for a given tumor type or have been intolerant to such therapy, or in the opinion of the Investigator have been considered ineligible for standard therapies on medical grounds, or refused to standard treatment (late or last line). Note: for subjects who are eligible based on intolerance to standard therapy or considered ineligible for standard therapies in the opinion of the investigator, the basis of this determination should be captured in the case report forms.
4. Willing to comply with the visits, study treatment, laboratory examinations and other study-related procedures and requirements specified in the study protocol.
5. Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
6. Expected survival time of more than 3 months.
7. Have at least one measurable lesion per RECIST version 1.1.
8. Adequate organ and bone marrow function:

   * Hematology (no blood transfusion, no G-CSF, no medication correction within 2 weeks prior to screening): Absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet (PLT) ≥ 100×109/L, hemoglobin (Hb) ≥ 90 g/L.
   * Liver function: total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 3.0×ULN, aspartate aminotransferase (AST) ≤ 3.0×ULN; for patients with liver metastases: ALT ≤ 5.0×ULN, AST ≤ 5.0×ULN;
   * Renal function: creatinine clearance (CrCL) ≥ 50 mL/min (calculated according to Cockcroft-Gault formula);
   * Coagulation function: prothrombin time (PT) ≤ 1.5×ULN or international normalized ratio (INR) ≤ 1.5×ULN, and activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
9. For female patients:

   * Females of childbearing potential who are not breastfeeding must agree to use highly effective contraceptives from the time of signing the ICF and use such contraceptives during the study and for at least 6 months after the last dose of the study drug; The blood pregnancy test result (human chorionic gonadotropin, hCG) must be negative within 3 days prior to enrollment.
   * Women who are infertile (i.e., physiologically incapable of becoming pregnant), including those surgically sterilized (having undergone bilateral oophorectomy, bilateral tubal ligation, or hysterectomy), or postmenopausal (non-treatment-induced amenorrhea) for ≥ 12 months prior to screening.
10. For male patients with fertile female partners, they must agree to use high-efficiency contraception from the time of signing the ICF and to use such contraception during the study and for at least 6 months after the last dose of the study drug.

Exclusion Criteria:

In order to participate in this study, all subjects must meet NONE of the exclusion criteria described.

1. Have received immune checkpoint inhibitors (ICIs) such as anti-PD-1 monoclonal antibody, anti-PD-L1 monoclonal antibody, anti-CTLA-4 monoclonal antibody, or VEGF inhibitor such as bevacizumab, ramucirumab, apatinib, or regorafenib within 28 days prior to the first dose of the study drug.
2. Known hypersensitivity to the study drug and any of its components; or known history of previous severe allergic reactions to macromolecular protein preparations/monoclonal antibodies or bispecific antibodies.
3. Female patient who is pregnant or breastfeeding.
4. Received major surgery within 4 weeks prior to the first dose of the study drug or requiring major elective surgery during the study period.
5. The adverse reactions caused by previous anti-tumor therapy have not been recovered to ≤ grade 1 per NCI CTCAE v5.0 (except for alopecia).
6. Subjects with untreated or symptomatic brain metastases, spinal cord compression, cancerous meningitis, or other evidence of uncontrolled brain or spinal cord metastases (Exception: Treated and stable symptoms, stable imaging for at least 4 weeks prior to first dose, with no evidence of cerebral edema, and no need for glucocorticoid therapy).
7. Patients with pleural effusion, pericardial effusion or ascites that have shown clinical symptoms or requiring repeated drainage.
8. Imaging during the screening period showed that the tumor surrounded important blood vessels or the presence of obvious tumor necrosis and cavitation, and the Investigator judged that entering the study may cause bleeding risk.
9. Known history of human immunodeficiency virus (HIV) infection (positive for HIV 1/2 antibody test) or diseases related to acquired immunodeficiency syndrome (AIDS).
10. Patients with hepatitis B infection undergoing treatment or requiring treatment (defined as hepatitis B surface antigen (HBsAg) positive, and HBV DNA >1000 copies/mL (200IU/mL) or above the lower limit of the detection, whichever is higher); or patients with hepatitis C antibody (HCV-Ab) positive and HCVRNA quantification > the upper limit of normal of the testing unit; or patients with known active syphilis infection.
11. Patients with uncontrolled bacterial, viral, fungal infections, or other pathogen infections (such as mycoplasma, parasites, etc.) that need systemic treatment within 4 weeks prior to the first dose of the study drug.
12. Known history of serious cardiovascular disease, including but not limited to:

    * Ventricular arrhythmia requiring clinical intervention.
    * Acute coronary syndrome (myocardial infarction and angina pectoris) within 6 months prior to the first dose of the study drug.
    * Congestive heart failure (New York Heart Association (NYHA) class ≥ II) or left ventricular ejection fraction (LVEF) < 50%;
    * QTc > 470 msec
    * Uncontrolled hypertension (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90 mmHg) after standard of care or poor compliance to antihypertensive therapy.
    * Major vascular disease (e.g., aortic aneurysm requiring surgery).
13. Patients with coagulation disorders, bleeding disorders, or other conditions having bleeding risk as judged by the Investigator, such as: skin wounds, surgical sites, trauma sites, mucosal severe ulcers or fractures that are not completely healed, or active gastroduodenal ulcer, intestinal obstruction, ulcerative colitis, esophagogastric varices, gastrointestinal perforation, etc. within 6 months before the first dose of the study drug.
14. Patients with ≥ grade 2 pulmonary hemorrhage/hemoptysis (according to NCI-CTCAE v5.0) within 1 month before the first dose of the study drug.
15. Patients with biopsy or other minor surgery within 7 days before the first dose of the study drug, except for placement of vascular access devices.
16. Patients experiencing arterial or venous thrombosis, stroke, or transient ischemic attack within 6 months before the first dose of the study drug.
17. Have received unstable doses of anticoagulant or thrombolytic drugs within 14 days of the first dose of the study drug. Please note that prophylactic use of low molecular weight heparin is allowed in the study.
18. Have received chronic treatment with aspirin (> 325 mg/day) or non-steroidal anti-inflammatory drugs known to inhibit platelet function; or received dipyridamole, ticlopidine, clopidogrel, or cilostazol within 14 days of first dose of the study drug.
19. Patients with diabetes mellitus poorly controlled by standard therapy (glycated hemoglobin HbA1c >8%).
20. Patients with current or past idiopathic pulmonary fibrosis or idiopathic pneumonia; current acute lung disease, interstitial lung disease or pneumonia (except for local interstitial pneumonia induced by radiotherapy), pulmonary fibrosis, etc.; Severe breathing difficulties, pulmonary insufficiency, or continuous oxygen inhalation.
21. Patients with active autoimmune disease, or history of autoimmune disease requiring systemic treatment within 2 years prior to screening, including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with the following conditions are eligible: hypothyroidism that can be controlled by hormone replacement therapy only, skin diseases (eg, vitiligo, psoriasis) that do not require systemic treatment, controlled celiac disease.
22. Received systemic corticosteroid treatment (prednisone > 10 mg/day or equivalent dose of similar drugs) or other systemic immunosuppressive treatment within 14 days before the first dose of the study drug.

    Patients with the following conditions are permitted: Treatment with topical, ocular, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; OR prophylactic short-term (≤ 7 days) use of corticosteroids (eg, hypersensitivity to contrast agent)); OR for the treatment of nonautoimmune diseases (such as delayed hypersensitivity reactions caused by contact allergens).
23. Received systemic antitumor therapy (chemotherapy, targeted therapy, biologic therapy, etc.) within 4 weeks or 5 half-lives (whichever is longer) before the first dose of study treatment; Received small molecule tyrosine kinase inhibitor therapy or hormonal antitumor therapy within 2 weeks before the first dose; received non-specific immunomodulatory therapy within 2 weeks before the first dose (such as interleukin, interferon, thymosin, cyclophosphamide, methotrexate, thalidomide, tumor necrosis factor, etc., excluding IL-11 for the treatment of thrombocytopenia); received Chinese herbal medicines or Chinese patent medicines with anti-tumor indications within 1 week before the first dose of the study drug.
24. For patients with hepatocellular carcinoma: Received locoregional treatment of the liver (such as transarterial chemoembolization, transcatheter embolization, hepatic arterial infusion, radiotherapy, radioembolization, or ablation) within 4 weeks prior to the first dose of the study drug.
25. Previously received organ or hematopoietic stem cell transplantation requiring the use of immunosuppressive agents.
26. History of other tumors within 5 years before screening, excluding skin basal cell carcinoma, skin squamous cell carcinoma, and cervical carcinoma in situ who underwent successful radical resection.
27. Received an attenuated vaccine within 4 weeks before screening or planned to receive an attenuated vaccine during the study.
28. Patients who participated in other clinical study and received other investigational agents or treatment within 4 weeks or 5 half-lives (whichever is longer) before the first dose of the study drug.
29. History of alcohol or drug abuse within 12 months prior to the first dose (for patients diagnosed with drug or alcohol abuse prior to 12 months prior to first dose, Enrollment only if no evidence of actual drug or alcohol abuse within 12 months prior to first dose).
30. Patient with any other medical or psychological condition, that is deemed by the Investigator to be likely to interfere with his/her ability to sign the informed consent, cooperate, or participate in the study.
31. Patients with other serious systemic diseases or conditions who are deemed unsuitable to participate in this clinical study at the judgement of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Escalation : DLT Assessment | From Day1 to Day15 after first dose of AP505
  Number of Participants With Dose Limiting Toxicity (DLT)
AE Assessment | From screening to follow-up period which includes safety follow-up (30/60/90 days after last dose) and survival follow-up (every 3 months until subject loss to follow-up, death, withdrawal of consent, or study termination, whichever occurs first).
  All AEs and SAEs will be collected, regardless of the relationship to the IP.
Determine the maximum tolerated dose (MTD) | From first dose of AP505 until 28 days after the last dose of AP505
Determine the recommended phase II dose (RP2D) | From first dose of AP505 until 28 days after the last dose of AP505

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile of AP505 in patients with advanced solid tumors | From C1D1 until 7 days after treatment discontinuation/ termination.
  Peak Plasma Concentration (Cmax) Analysis
To evaluate the pharmacokinetic (PK) profile of AP505 in patients with advanced solid tumors | From first dose until 7 days after treatment discontinuation/ termination.
  Area under the plasma concentration versus time curve (AUC) Analysis
To evaluate the pharmacokinetic (PK) profile of AP505 in patients with advanced solid tumors | From first dose until 7 days after treatment discontinuation/ termination.
  Terminal elimination half-life (t1/2) Analysis
To evaluate the pharmacokinetic (PK) profile of AP505 in patients with advanced solid tumors | From first dose until 7 days after treatment discontinuation/ termination
  Time to reach the maximum observed concentration (Tmax) Analysis
To characterize the immunogenicity profile of AP505 in patients with advanced solid tumors | From C1D1 (Cycle 1 is 15 days ; Cycle 2 onwards: each cycle is 28 days), until safety follow up (up to 90 days after the last dose).
  Immunogenicity indicators: the level of anti-drug antibody (ADA).
To characterize the immunogenicity profile of AP505 in patients with advanced solid tumors | From C1D1 (Cycle 1 is 15 days ; Cycle 2 onwards: each cycle is 28 days), until safety follow up (up to 90 days after the last dose).
  Immunogenicity indicators: the level of NAb (if ADA is positive).

CONTACTS AND LOCATIONS:
Locations (1):
- AP Biosciences, Inc., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No